CLINICAL TRIAL: NCT06689657
Title: Randomized Study of Two Modalities of Cognitive-behavioral Group Therapy in Adolescents with Suicidal Ideation or Suicidal Behavior
Brief Title: Understanding and Acting to Regulate Suicidal Behavior
Acronym: CARES
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: RECHMPL22_0339 / UF 8379
Record Dates: First submitted 2024-11-13; First posted 2024-11-14 (Actual); Last update posted 2024-11-14 (Actual); Status verified 2024-11

CONDITIONS: Suicidal Ideation; Suicidal Behavior; Self-harm Behavior; Adolescents
Keywords: Suicide prevention; Cognitive-behavioral therapy; Dialectical Behavior Therapy; Non pharmacological intervention; Adolescent
MeSH Terms: conditions — Suicidal Ideation; Suicide Prevention

STUDY DESIGN:
Intervention Model Description: Adolescent group therapy (CARES) and parent group therapy (RNV) vs Adolescent groupe therapy (CARES) only
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Adolescent group therapy (CARES) and parent group therapy (RNV) (Other): In the adolescent group, they will attend 8 group sessions during 1 month (2 sessions/week). There also will be a "boost" session 3 month after the last session.
  Parents will attend 4 group sessions during 1 month too (1 session/week). There will be 2 "boost" sessions : 1 month and 3 month after the last session
  Patients will be randomized in each group with blinded assessment
  Interventions: Other: Adolescent group therapy (CARES) and parent group therapy (RNV)
- Adolescent groupe therapy (CARES) only (Experimental): In the adolescent group, they will attend 8 group sessions during 1 month (2 sessions/week).
  There will be a "boost" session 3 month after the last session
  Patients will be randomized in each group with blinded assessment
  Interventions: Behavioral: Cognitive behavioral group therapy for adolescents and non violent resistance group for parents

INTERVENTIONS:
Behavioral: Cognitive behavioral group therapy for adolescents and non violent resistance group for parents — In the adolescents group, this cognitive-behavioral group therapy will include emotion regulation skills, distress tolerance skills, cognitive strategies, work on values and problem-solving strategies
  Those sessions will include psychoeducation about adolescents, about suicidal ideation and suicidal behavior, coping with adolescent emotional distress, support on how to be a parent today (screen regulation...) and manage daily life
  Arms: Adolescent groupe therapy (CARES) only
Other: Adolescent group therapy (CARES) and parent group therapy (RNV) — In the adolescent group, they will attend 8 group sessions during 1 month (2 sessions/week). There also will be a "boost" session 3 month after the last session. Parents will attend 4 group sessions during 1 month too (1 session/week). There will be 2 "boost" sessions : 1 month and 3 month after the last session Patients will be randomized in each group with blinded assessment
  Arms: Adolescent group therapy (CARES) and parent group therapy (RNV)

SUMMARY:
Data from Santé Publique France show that since the onset of the health crisis (covid-19), there has been an increase in emergency room visits for mood disorders among children under 15 years of age, with a notable rise in the number of visits since early September 2020 compared to previous years. Recent literature considers Dialectical Behavior Therapy (DBT) as the only approach that has demonstrated (albeit weak to moderate) effects on the recurrence of self-harming behaviors. It is within this context, and based on these various findings, that the CARES program was developed (Understanding and Acting to Regulate Emotions and Suicidal Behaviors), aimed at adolescents who have engaged in suicidal behaviors or who have active suicidal ideation.

The objective of this study is to compare the CARES program for adolescents alone to the CARES program for adolescents combined with a parent group using Non-Violent Resistance (NVR) on the occurrence of self-harming behaviors among adolescents who have engaged in suicidal acts and/or have active suicidal ideation, six months after the conclusion of the intervention.

This is a prospective, randomized, open-label, single-center, controlled study with two parallel arms, with blinded assessment of the outcome measures.

DETAILED DESCRIPTION:
The CARES adolescent program consists of a group intervention with 8 biweekly sessions over a total duration of one month, followed by a booster session 3 months post-intervention. These sessions are conducted by nurses and psychologists trained in Cognitive Behavioral Therapies (CBT). The content of the group aims to provide adolescents with cognitive and behavioral strategies to improve their emotional distress tolerance and to expand their repertoire of solutions in times of emotional crisis.

The CARES adolescent and NVR parent program includes the same adolescent group described above, supplemented by an NVR parent group. This parent group meets once a week for one month (4 sessions), with two additional booster sessions at 1 month and 3 months post-intervention. The content of the parent program is a parent management training composed of strategies for managing their adolescent's emotional crises through emotional regulation techniques based on Non-Violent Resistance (NVR) methods (Omer, 2021).

ELIGIBILITY:
Inclusion Criteria:

* Age from 12 to 16 years 11 months old
* Active suicidal ideation and/or suicidal behavior during the last 6 months
* The patient is referred by a healthcare professional

Exclusion Criteria:

* Intellectual developmental disorder
* Non-french speaking
* Planned travel not allowing the complete following of the study
* The patient, the parents or the legal guardian can not be correctly informed
* The patient presents symptoms that prevent him from group interaction (behavior disorders, hallucinations, delirium)
* The family already followed the same kind of program
* The patient is already enrolled in a clinical trial or is taking a treatment off full market approval during 4 weeks before screening
* The patient and the family are not affiliated to any healthcare insurance
* No signed consent from parents or a legual guardian nor one of the parental authority holder
* The patient did not consent

Ages: 12 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 108 (Estimated)
Dates: Start 2025-01-06 (Estimated); Primary Completion 2028-01-06 (Estimated); Study Completion 2028-07-06 (Estimated)

PRIMARY OUTCOMES:
Occurence of suicidal behavior | Variation between initial assessment and assessment 6 month post intervention
  Assessed with the Columbia Suicide Severity Rating Scale (C-SSRS)

SECONDARY OUTCOMES:
Clinical improvement assessement (clinician) | Variation between initial assessment and post-intervention and between initial assessment and 6 months post-intervention
  Assessment with the Clinical Global Impression-Improvement (CGI-I)
Parenting stress | Variation between initial assessment and post-intervention and between initial assessment and 6 months post-intervention
  Assessment with the Parenting Stress Index short form (PSI-4-SF)
Parenting anxiety and depression | Variation between initial assessment and post-intervention and between initial assessment and 6 months post-intervention
  Assessment with the Hospital Anxiety and Depression Scale (HADS)
Adolescent depression | Variation between initial assessment and post-intervention and between initial assessment and 6 months post-intervention
  Assessment with the Child Depression Inventory (CDI)
Suicidal ideation | Variation between initial assessment and post-intervention and between initial assessment and 6 months post-intervention
  Assessment with the C-SSRS